CLINICAL TRIAL: NCT05461014
Title: Evaluating the Acceptability, Feasibility Utilization of a Digital Behavioral Tool for Adolescents and Young Adults With IBD Who Are in the Process of Transitioning From Pediatric to Adult Care
Brief Title: RxWell in Pediatric IBD for Disease Management and Transition Readiness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sandra Kim, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21100037
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Mental Health Issue; Inflammatory Bowel Diseases
Keywords: mobile app; digital behavioral tool; adolescent and young adult
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Cognitive Behavioral Intervention (DCBI) (Experimental): The dCBI, RxWell, is a trans cognitive behavioral therapy (CBT) mobile app product addressing depression and anxiety that was developed based on standard CBT techniques.
  Interventions: Behavioral: dCBI

INTERVENTIONS:
Behavioral: dCBI — The dCBI, RxWell, is a trans-CBT mobile app product addressing depression and anxiety that was developed based on standard CBT techniques. RxWell provides users users with 40 brief (5-10 minute) skill building techniques for anxiety and depression. Users will have access to a goal-setting tab and "in the moment relief" section which contains over 17 techniques,14 of which are brief audios to help users engage relaxation responses. The user will be provided with the depression path, which has 40 unique techniques, and if the user expresses significant anxiety, the coach will have the ability to personalize the program by pulling in any of the 53 techniques from the anxiety path, so that the individual can utilize the proper CBT techniques that fit with their presentation. The coaches are trained to provide assistance with adult care transition readiness.

SUMMARY:
Evaluate the feasibility and acceptability of adapted coached RxWell for patients ages 16-25. Adapt and beta test the modified RxWell product to include chronic disease management and transition readiness. Evaluate RxWell usage and its impact to the TRAQ questionnaire over time.

DETAILED DESCRIPTION:
Baseline TRAQ and PHQ-4 scores will be obtained from the patient as part of routine care during annual visits or as a screening tool after consent to determine eligibility. If the patient is recruited from a visit other than the annual visit, the TRAQ and PHQ4 will be completed to determine eligibility after consent. If eligible, the participant will complete the IBD self-efficacy scale, GAD7, and PHQ8, and will be provided with an access code to download RxWell and will be paired with a UPMC digital health coach who will guide the person through the sessions and text within the app to help give them the tools needed to actively cope with anxiety and/or depression. The adapted version of RxWell includes the same RxWell content/techniques but the coaching model within the adapted version has increased responsibilities of the coach, encouraging the development of necessary transition knowledge and skills for the patient. Coaches in this version will also participate in training about how best to interact with IBD patients regarding their chronic illness, transitions to adult physician, and care management. These coaches will be supervised by a licensed UPMC mental health clinician. The coaches will be informed of the reason for each user's access to the dCBI, TRAQ or PHQ score or both and will interact with the user accordingly. Participants will be asked to complete all study measures (TRAQ, PHQ8, IBD Self-Efficacy, and GAD7) at all time points, baseline, 3 and 6 months.

The user will have access to the app and coach for six months after they have consented. Each technique that is used during those six months will be stored in the practice-again section and available to the participant for use during the study. After six months, participants will no longer have access to the app and will be informed about this change. Participants are informed when they sign up for this app that is not a crisis management tool. There is a risk escalation protocol in place at UPMC if the content of patient's messaging to coaches is alarming.

A randomly selected group of patients who consent to this study and engage with the app, meaning completing 3 or more techniques and/ or actively engaged with the coach, will participate in qualitative interviews to determine how to best implement disease self-management tools within the digital behavioral tool. Every third participant who consents and meets the engagement criteria will be contacted to complete the qualitative interview.

All participants will also be asked to complete quantitative assessments at baseline and again 3 and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 16-25 years with established IBD who are followed in the pediatric gastroenterology clinics at the UPMC Children's Hospital of Pittsburgh
* Patient must be English speaking
* Access to Smartphone
* PHQ-4 score ≥ 5 and/or TRAQ score ≥ 60

Exclusion Criteria:

* Developmental delay

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Change in anxiety severity over time | 6 months
  Generalized Anxiety Disorder 7 measures anxiety severity (score ranges from 0-21, with 21 being severe anxiety) is completed within the app and at three study timepoints (baseline, 3 months and 6 months). This measure will be studied over time, up to 6 months.
Change in depression severity | 6 months
  Patient Health Questionnaire 8 to measures depression severity (score ranges from 0-24, with 24 being severe depression) is completed within the app and at three study timepoints (baseline, 3 months and 6 months). This measure will be studied over time, up to 6 months.

SECONDARY OUTCOMES:
Change in Transition Readiness to Adult Care | 6 months
  Change in transition readiness assessment questionnaire that measures the readiness of a patient to care for their own medical needs without parental/guardian support (score ranges from 20-100 where the higher score demonstrates higher competency in caring for one's own needs) is completed at baseline, 3 and 6 months. This measure will be studied over time, up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Kim, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. Data will be shared at the aggregate level.